CLINICAL TRIAL: NCT05110365
Title: Effects of Proprioceptive Neuromuscular Facilitation Exercise on Blood Pressure and Ankle Brachial Index in Patient With Hypertension
Brief Title: Effect of Proprioceptive Neuromuscular Facilitation on Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/01045 Raja Saddam
Record Dates: First submitted 2021-10-26; First posted 2021-11-05 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Hypertension
Keywords: proprioceptive neuromuscular facilitations; ankle brachial index; diabetes
MeSH Terms: conditions — Hypertension; Diabetes Mellitus | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- proprioceptive neuromuscular facilitation (Experimental): proprioceptive neuromuscular facilitation techniques
  Interventions: Other: Proprioceptive Neuromuscular Facilitation
- control (No Intervention): no intervention

INTERVENTIONS:
Other: Proprioceptive Neuromuscular Facilitation — The patient will be provided with mild to moderate resistance PNF pattern which is a type of Endurance training which decreases BP through a reduction in systemic vascular resistance(15).In a regimen as follow with the frequency of 3 days a week, a repetition of 3 sets for one hour and a total duration of 3 months(16). The PNF patterns will be diagonal 1 (D1) and diagonal 2 (D2) patterns. Both patterns are subdivided into: A) Moving into Flexion: the toes start flexed and ends extended. Ankle and foot start plantar flexed; everted and ends dorsiflexed inverted. Tibia starts externally rotated and ends internally rotated. Knee starts extended, and ends flexed. The hip starts extended, abducted, internally rotated and ends flexed, adducted, externally rotated.B) Moving into Extension: The start and end are reversed to "D1 Moving into Flexion"
  Arms: proprioceptive neuromuscular facilitation

SUMMARY:
To determine the effect of Proprioceptive Neuromuscular Facilitation exercise on blood pressure in patient with mild to moderate hypertension.Both genders will be included.Patients aged between 40 and 60 years with mild and moderate hypertension.Systolic blood pressure 130-160 mmHg or Diastolic Blood Pressure 80-100 mmHg.

Sphygmomanometer and EuroQoL five-dimensional instrument would be used for the 'Pre' & 'Post' assessment.

DETAILED DESCRIPTION:
There is a belief that proprioceptive neuromuscular facilitation exercises cause cardiac overload as blood pressure in immediately influenced by exercise but Pereira concluded in his research that proprioceptive neuromuscular facilitation exercises with minimum repetitions are safe for hypertensive or cardiovascular patients because in his study there is no increase in blood pressure in older women after performing three different types of PNF exercises. Pereira discovered that rhythmic initiation , dynamic reversals , and combination of isotonic techniques did not raise blood pressure levels, thus it is recommended to use up to five repeats of repetition maximum . One study observed at the effects of passive and modified proprioceptive neuromuscular facilitation (PNF)stretching techniques on acute systolic and diastolic blood pressure responses. All PNF treatments were beneficial in increasing Range of motion, as we all know.

PNF improves Range Of Motion while avoiding an increase in Systolic blood pressure in one or two trials, but increases Systolic blood pressure in a third trial. Blood pressure rises by 40% with conventional exercise programmers and because PNF involves near-maximal resistance,researchers anticipated a considerable rise in blood pressure during PNF execution. It was discovered that elderly subjects could not readily execute more than five to seven repetitions of PNF exercises, which has also been shown by others. Due to the low repetition number of each movement pattern, the results showed that PNF did not induce a high enough workload to increase blood pressure in the elderly.

ELIGIBILITY:
Inclusion Criteria:

* Both genders will be included.
* Patients aged between 40 and 60 years with mild and moderate hypertension.
* Systolic blood pressure 130-160 mmHg or Diastolic blood pressure 80-100 mmHg.
* Mild and moderate hypertension with diabetes

Exclusion Criteria:

* Severe hypertensive patients.
* Patient on smoking
* Patient with severe complications and comorbidities.
* Not willing to give consent/ data

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-06-26 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-08-18 (Actual)

PRIMARY OUTCOMES:
sphygmomanometer | 12 weeks
  sphygmomanometer will be used for measuring blood pressure and ankle brachial index

SECONDARY OUTCOMES:
(EuroQoL five-dimensional instrument ) | 12 weeks
  quality of life measures the five dimension mobility,selfcare,usual activities,pain and anxiety.
  0 for minimum 5 for maximum

CONTACTS AND LOCATIONS:
Overall Officials: sania aziz, MSNMPT, Principal Investigator — Riphah International University
Locations (1):
- Valley Medical Complex Abbottabad, Abbottābād, Kpk, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Linke A, Erbs S, Hambrecht R. Effects of exercise training upon endothelial function in patients with cardiovascular disease. Front Biosci. 2008 Jan 1;13:424-32. doi: 10.2741/2689. PMID 17981557
- [Background] Papaioannou TG, Oikonomou E, Lazaros G, Christoforatou E, Vogiatzi G, Tsalamandris S, Chasikidis C, Kalambogias A, Mavratzas T, Stofa E, Mystakidi VC, Latsios G, Deftereos S, Tousoulis D. Arterial stiffness and subclinical aortic damage of reclassified subjects as stage 1 hypertension according to the new 2017 ACC/AHA blood pressure guidelines. Vasa. 2019 May;48(3):236-243. doi: 10.1024/0301-1526/a000765. Epub 2018 Dec 10. PMID 30526401
- [Background] Varounis C, Katsi V, Nihoyannopoulos P, Lekakis J, Tousoulis D. Cardiovascular Hypertensive Crisis: Recent Evidence and Review of the Literature. Front Cardiovasc Med. 2017 Jan 10;3:51. doi: 10.3389/fcvm.2016.00051. eCollection 2016. PMID 28119918
- [Background] Singh S, Shankar R, Singh GP. Prevalence and Associated Risk Factors of Hypertension: A Cross-Sectional Study in Urban Varanasi. Int J Hypertens. 2017;2017:5491838. doi: 10.1155/2017/5491838. Epub 2017 Dec 3. PMID 29348933
- [Background] Papadopoulos DP, Sanidas EA, Viniou NA, Gennimata V, Chantziara V, Barbetseas I, Makris TK. Cardiovascular hypertensive emergencies. Curr Hypertens Rep. 2015 Feb;17(2):5. doi: 10.1007/s11906-014-0515-z. PMID 25620633
- [Background] Hindle KB, Whitcomb TJ, Briggs WO, Hong J. Proprioceptive Neuromuscular Facilitation (PNF): Its Mechanisms and Effects on Range of Motion and Muscular Function. J Hum Kinet. 2012 Mar;31:105-13. doi: 10.2478/v10078-012-0011-y. Epub 2012 Apr 3. PMID 23487249
- [Background] Kim EK, Lee DK, Kim YM. Effects of aquatic PNF lower extremity patterns on balance and ADL of stroke patients. J Phys Ther Sci. 2015 Jan;27(1):213-5. doi: 10.1589/jpts.27.213. Epub 2015 Jan 9. PMID 25642076
- [Background] Pereira MP. Proprioceptive neuromuscular facilitation does not increase blood pressure of healthy elderly women. Physiother Theory Pract. 2012 Jul;28(5):412-6. doi: 10.3109/09593985.2011.609582. Epub 2011 Oct 18. PMID 22007735
- [Background] Fagard RH, Cornelissen VA. Effect of exercise on blood pressure control in hypertensive patients. Eur J Cardiovasc Prev Rehabil. 2007 Feb;14(1):12-7. doi: 10.1097/HJR.0b013e3280128bbb. PMID 17301622